CLINICAL TRIAL: NCT07075861
Title: JenaValve Trilogy for Patients With Pure Native Aortic Valve Rigurgitation: the ARTEMIS Data Collection Study
Brief Title: The ARTEMIS Data Collection Study
Acronym: ARTEMIS
Status: Recruiting | Type: Observational
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Sponsor
Other Study IDs: CET 203-2025
Record Dates: First submitted 2025-07-10; First posted 2025-07-20 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-11

CONDITIONS: Aortic Regurgitation Disease
Keywords: JenaValve Trilogy; Aortic Regurgitation; TAVI
MeSH Terms: conditions — Aortic Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with symptomatic, severe, native aortic regurgitation: patients with symptomatic, severe, native aortic regurgitation retrospectively or prospectively treated with TAVI JenaValve

SUMMARY:
To observe the safety and effectiveness of the JenaValve Trilogy™ Heart Valve System for transcatheter aortic valve replacement (TAVR) in subjects with evere native aortic regurgitation (AR) who are indicated for TAVR Data collection

DETAILED DESCRIPTION:
To observe the safety and effectiveness of the JenaValve Trilogy™ Heart Valve System for transcatheter aortic valve replacement (TAVR) in subjects with evere native aortic regurgitation (AR) who are indicated for TAVR Data collection .

A retrospective/prospective, single-arm, post-market study to monitor the outcomes of Jena Valve Trilogy in a real-world clinical setting .

After enrollment is completed, patients are followed to 1 year (an amendment to extend the follow up to 5 years will be evaluated). Thereafter, the patient exits the data collection study and is to be followed per institutional standard of care for TAVR patients.

The JenaValve Trilogy™ Heart Valve System contains the following sub-components: a prosthetic transcatheter porcine pericardial aortic valve, 20Fr Introducer Sheath System, transfemoral Delivery Catheter, and Loading Tool.

Indications for Use: The JenaValve Trilogy™ Heart Valve System is indicated for use in patients with clinically significant aortic regurgitation (AR) who are considered high risk candidates for surgical aortic valve replacement as deemed by the local multi-disciplinary heart team.

This is an investigator initiated study that will include 75 suitable patients according to the inclusion/exclusion criteria as per IFU.

ELIGIBILITY:
Inclusion Criteria:

* Considered at high or prohibitive risk for surgical aortic valve replacement by the Heart Team

  * 18 years of age or older
  * Suitable anatomy according to the IFU
  * Absence of significant disease of the ascending aorta, including ascending aortic aneurysm (defined as maximal luminal diameter of 50mm or greater) or atheroma (especially if thick [>5mm], protruding or ulcerated)

Exclusion Criteria:

The JenaValve Trilogy Heart Valve System is contraindicated for use in patients who have known hypersensitivity or contraindication to Nitinol (titanium and/or nickel), an anti-coagulation/anti-platelet regimen or contrast medium that cannot be managed with premedication, or who have active bacterial endocarditis or other active infections.

The JenaValve Trilogy Heart Valve System is contraindicated in those patients whose anatomy does not accommodate the System due to anatomical considerations outlined in the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with severe symptomatic aortic valve regurgitation in a native valve. According to the local experience in TAVR, the number of patients with severe AR deemed at prohibitive surgical risk is around 2/month. Considering a prospective enrollment of 2 years and historical patients collected data for 1 year, the final number of expected patients will be about 75. In fact, according to reference [1], a composite of all-cause mortality and heart failure ehospitalization at 1 year had cumulative incidence of about 17%. Therefore, considering an exponential distribution with event rate 0.17 (17 events per 100 person years), 75 patients amount to a total of 75-13*.5=68 person years. The resulting 95% confidence interval of the cumulative incidence will be 0.06; 0.24 [2].
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2025-08-10 (Actual); Primary Completion 2028-08-10 (Estimated); Study Completion 2028-08-10 (Estimated)

PRIMARY OUTCOMES:
Device success at 12 months | 12 months
  Freedom from all-cause mortality
  * Freedom from unsuccessful delivery of the device, and retrieval of the delivery system
  * Freedom from incorrect positioning of a single prosthetic heart valve into the proper anatomical location
  * Freedom from surgery or intervention related to the device or to a major vascular or access-related or cardiac structural complication
  * Intended performance of the valve (i.e., no moderate or severe prosthetic valve regurgitation)

CONTACTS AND LOCATIONS:
Overall Officials: Luca Testa, PI, Principal Investigator — IRCCS Policlinico San Donato (San Donato Milanese) - IT
Locations (1):
- IRCCS Policlinico San Donato, San Donato Milanese, Milano, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-04-15): https://cdn.clinicaltrials.gov/large-docs/61/NCT07075861/Prot_SAP_002.pdf
  • Informed Consent Form (2025-04-15): https://cdn.clinicaltrials.gov/large-docs/61/NCT07075861/ICF_001.pdf